CLINICAL TRIAL: NCT04571164
Title: A Multi-centre,Randomized,Double-blind,Placebo Parallel Controlled Study to Evaluate the Effectiveness and Safety of LY03003 in Patients With Early Primary PD
Brief Title: A Study to Evaluate the Effectiveness and Safety of LY03003 in Patients With Early Primary PD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Luye Pharma Group Ltd. (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LY03003/CT-CHN-304
Record Dates: First submitted 2020-09-21; First posted 2020-09-30 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Parkinson Disease
Keywords: parkinson disease; LY03003
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LY03003 (Experimental)
  Interventions: Drug: LY03003(Rotigotine,extended-release microspheres)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo,extended-release microspheres

INTERVENTIONS:
Drug: LY03003(Rotigotine,extended-release microspheres) — During the intervention, the initial dose was 14mg, and then was incremented in weekly units, 14mg each time, until the maximum dose of 56mg set in this study was reached 4 weeks after titration, the optimal therapeutic dose or the maximum tolerated dose was entered into the dosing maintenance period. After entering the maintenance period, no dose adjustment was performed, and the stable dose was maintained for 24 weeks
  Arms: LY03003
Drug: Placebo,extended-release microspheres — During the intervention,the initial does was 14mg,and then was incremented in weekly units,14mg each time,until the maximum does of 56mg set in this study was reached 4 weeks after titration,the optimal therapeutic does or the maximum tolerated does was entered into the dosing maintenance period.After entering the maintenance period,no does adjustment was performed,and the stable does was maintained for 24 weeks.
  Arms: Placebo

SUMMARY:
This study is to evaluate the effictiveness and safety of Ly03003 following intramuscular injections

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent must be given to the trial and written informed consent must be voluntarily signed, good communication with the investigator and compliance with all requirements of the clinical trial (planned visits, laboratory tests and other procedures);
2. Age ≥30 years old, regardless of gender;
3. The subject has had primary Parkinson's disease for less than 5 years, and the diagnosis is based on the main symptom -- motor delay plus at least 1 symptom: quiescence tremor, myotonia, and no other known or suspected cause of Parkinson's disease;
4. Hoehn-yahr grading ≤3 (excluding 0);
5. Brief mental state examination (MMSE) ≥25 points;
6. Unified Parkinson disease rating scale (UPDRS) motor score (part Ⅲ) 10 or higher;
7. If the subjects are receiving anticholinergic drugs (such as benzalkonium tropic, benzene hai suo, diethyl promethazine, its organism and than pp board), MAO - B inhibitors (e.g., company to gillan, LeiSha gillan), NMDA antagonists, such as amantadine treatment, must dose before baseline stability at least 28 days, and maintain the dose treatment during the study period
8. Women of childbearing age (defined as women who have not undergone surgical sterilization or less than 1 year after menopause) or male subjects agree to use reliable contraceptives (oral contraceptives, condom use, abstinence, etc.) throughout the study period (until the end of the study), and pregnancy outcomes were negative for women of childbearing age at screening and baseline.

Exclusion Criteria:

1. History of pallidotomy, thalamotomy, deep brain stimulation or fetal tissue transplantation
2. Dementia, active mental illness or hallucination, major depression
3. Those who received dopamine receptor agonists within 28 days before baseline
4. Patients receiving levodopa preparation (including levodopa compound preparation) within 28 days before baseline, or levodopa preparation after diagnosis for more than 6 months
5. Patients receiving any of the following drugs within 28 days before baseline: amphetamine, metoclopramide, α-methyldopa, antipsychotics, MAO-Ainhibitors, flunarizine, reserpine, methylphenidate, budesonide, etc
6. Active central nervous system drugs (such as sedatives, hypnotics, antidepressants, and antianxiety drugs) are under treatment, except those who have maintained a stable dose for at least 28 days before the baseline (visit 2) and may remain stable during the study period
7. Atypical Parkinson's disease symptoms caused by taking drugs (such as metoclopramide, flunarizine), hereditary metabolic diseases of nervous system (such as Wilson's disease), encephalitis, cerebrovascular diseases or degenerative diseases (such as progressive supranuclear paralysis)
8. Have a history of epilepsy, or have a history of stroke or transient cerebral ischemia within 1 year before the visit
9. Those who are intolerant or allergic to the following antiemetic drugs, such as domperidone, trimethoxybenzamide, ondansetron, tropisetron, granisetron and glinbromide
10. Patients with clinically significant abnormal liver function were defined as total bilirubin > 1.5 times of the upper limit of the reference value range or ALT or ast > 2 times of the upper limit of the reference value range
11. Patients with clinically significant renal dysfunction (serum creatinine > 2.0 mg / dl [> 177 μ mol / l])
12. Patients with uncontrollable or important cardiovascular diseases, including congestive heart failure of NYHA grade II or above, unstable angina pectoris, myocardial infarction within 6 months before the first administration of trial drug, or arrhythmia requiring treatment at the time of screening
13. At screening, QTc interval: male > 450ms, female > 460ms
14. Patients with a history of orthostatic hypotension, or those with SBP ≥ 20mmhg or DBP ≥ 10mmhg at screening (visit 1) and baseline (visit 2) when switching from supine position to upright position for 1 or 3 minutes; or those with SBP < 105mmhg at visit 1 and visit 2;
15. Subjects with evidence of impulse control disorder (ICD) during screening (visit 1);
16. A history of suicide attempt (including actual attempt, interruption or failure of attempt) or suicidal ideation in the past 6 months were defined as those who answered "yes" to question 4 or question 5 of the Columbia suicide severity rating scale (c-ssrs) during screening (visit 1);
17. Patients with history of narcolepsy;
18. Those who had a history of alcoholism, drug abuse and drug abuse in the past five years (visit 1) were screened. Alcoholism was defined as drinking more than 14 units of alcohol per week (1 unit = 360 ml beer or 45 ml alcohol with 40% alcohol content or 150 ml wine);
19. Patients with malignant tumor within 5 years before screening were excluded from cervical carcinoma in situ, skin basal cell or squamous cell carcinoma, local prostate cancer after radical operation and breast intraductal carcinoma in situ after radical operation;
20. Pregnant or lactating women;
21. The patients who had participated in the rotigotine test were intolerable or ineffective;
22. Allergic constitution (allergic to two or more drugs or foods) or known to be allergic to rotigotine or rotigotine microspheres;
23. Those who have participated in clinical trials of other drugs within 3 months before screening;
24. Other clinically significant medical status, mental status or laboratory abnormalities judged by the researcher may interfere with the subject's ability to participate in the study.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 294 (Actual)
Dates: Start 2020-05-11 (Actual); Primary Completion 2022-03-17 (Actual); Study Completion 2022-09-27 (Actual)

PRIMARY OUTCOMES:
Change from baseline to the end of the treatment period in the Unified Parkinson's Disease Rating Scale(UPDRS)part(Ⅱ+Ⅲ)Total Score | From baseline to the end of the double-blind dose maintenance period at 24weeks

SECONDARY OUTCOMES:
The proportion of patients whose total UPDRS decreased by 20、25、30percent or mors | From baseline to the end of the double-blind dose maintenance period at 24weeks
UPDRS scale part Ⅱchanges relative to the baseline | From baseline to the end of the double-blind dose maintenance period at 24weeks
UPDRS scale part Ⅲchanges relative to the baseline | From baseline to the end of the double-blind dose maintenance period at 24weeks
Changes in SI scores in the Total Clinical Efficacy Rating Scale (CGI) relative to baseline,the scores of GI and EI | From baseline to the end of the double-blind dose maintenance period at 24weeks
To clarify the changes in PDQ-8 questionnaire scores relative to baseline | From baseline to the end of the double-blind dose maintenance period at 24weeks
To clarify the changes in PDSS questionnaire scores relative to baseline | From baseline to the end of the double-blind dose maintenance period at 24weeks
To clarify the changes in BDI-Ⅱquestionnaire scores relative to baseline | From baseline to the end of the double-blind dose maintenance period at 24weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital Capital Medical University, Beijing, China